CLINICAL TRIAL: NCT07300826
Title: Intravenous Dexmedetomidine Versus Midazolam in Preventing Shivering in Trauma Patients Undergoing Lower Limb Orthopedic Surgery Under Spinal Anesthesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Gad, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dexmedetomidine VS Midazolam
Record Dates: First submitted 2025-12-20; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lower Limb Orthopedic Surgery
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group D (Experimental): Patients will receive i. v. dexmedetomidine 0.5 μg.kg-1 post-spinal anesthesia
  Interventions: Drug: Dexmedetomidine
- Group M (Experimental): and patients will receive i.v. midazolam 0.05 mg.kg-1 post-spinal anesthesia
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive i. v. dexmedetomidine 0.5 μg.kg-1 post-spinal anesthesia
  Arms: Group D
Drug: Midazolam — patients will receive i.v. midazolam 0.05 mg.kg-1 post-spinal anesthesia
  Arms: Group M

SUMMARY:
Shivering is a common and significant complication following spinal anesthesia, with a reported incidence of 40-60% especially in trauma patients due to pain, stress response, blood loss, and disrupted thermoregulation. Shivering increases oxygen demand, impairs monitoring, and reduces patient comfort. Effective pharmacologic prevention of shivering is crucial in this population.

Dexmedetomidine is a highly selective α2-adrenoreceptor agonist. It is widely used as an adjunct to general as well as regional anesthesia for better hemodynamic stability, sedation, and prolonged duration of regional anesthesia and is effective in reducing shivering by centrally modulating thermoregulation.

Midazolam, a GABA-A agonist, Intravenous midazolam premedication is commonly used for conscious sedation, anxiolysis, and amnesia with spinal anesthesia is also known to have anti-shivering properties attributed to its action on GABA-A receptors, promoting anxiolysis and possibly resetting the hypothalamic thermoregulatory threshold.

There are limited clinical data comparing the effect of intravenous dexmedetomidine and midazolam and its effect on shivering

ELIGIBILITY:
Inclusion Criteria:

* : ASA I-II Adult trauma patients (age 18-60 years). Undergoing lower limb orthopedic surgery with tourniquet under spinal anesthesia

Exclusion Criteria:

- Allergy to study drugs. Severe cardiovascular, hepatic, or renal disease Hypovolemic shock. History of psychiatric illness or chronic sedative use. Bradycardia (<50 bpm), heart block, or uncontrolled hypotension. Febrile illness or use of active warming devices

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of shivering | 1 hours postoperative
  Incidence of shivering intraoperatively every 10 min and postoperatively every 15 min for 1 hour